CLINICAL TRIAL: NCT06859242
Title: Development and Validation of a Risk Prediction Model for Iodinated Contrast Medium Extravasation in Patients Undergoing Contrast-enhanced Computed Tomography
Brief Title: Risk Prediction Model for Iodinated Contrast Medium Extravasation
Acronym: RPMICME
Status: Recruiting | Type: Observational
Sponsor: Zhang Wenyan (Other)
Responsible Party: Sponsor-Investigator, Zhang Wenyan, Principle Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: myanna2010; 2024D24 (Other Grant/Funding Number: TongjiHospital)
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Extravasation of Contrast Media
Keywords: Extravasation of Contrast Media; Predictive Models; Machine; Risk Management
MeSH Terms: conditions — Extravasation of Diagnostic and Therapeutic Materials

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop a risk prediction model for iodine contrast agent extravasation from peripheral veins and to implement this model clinically to establish a risk control management system for iodine contrast agent extravasation.A case-control study design was employed to collect data for model development. The case group comprised patients who experienced iodine contrast agent extravasation during enhanced CT examinations, while the control group included patients who underwent similar examinations without extravasation.

DETAILED DESCRIPTION:
In this study, a retrospective case-control design was utilized to collect data from patients who underwent enhanced CT examinations at our medical center. In line with the nursing management protocols of our center, all cases of iodine contrast extravasation require treatment and follow-up, necessitating the creation of an electronic record for each affected patient. During the establishment of these records, researchers obtained consent from the affected patients to include them in the study. Upon receiving approval, relevant data from the records were extracted for research purposes. For the non-extravasation group, researchers approached eligible patients or their guardians after the examination, explained the study's objectives, and collected pertinent data through Electronic Medical Record System after obtaining informed consent.

The collected data encompass general demographic information (including age, gender, height, and weight), medical history (including conditions such as malignant tumors, chemotherapy treatments, hypertension, and diabetes), and examination parameters (including specific examination items, types of contrast agents, injection dosages, and flow rates). Additionally, the dataset includes venous access details (such as vascular conditions, peripheral venous catheter insertion sites, and catheter models) and environmental factors (such as maximum and minimum temperatures and temperature variations).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in this study.
2. Without contraindications such as iodine contrast allergy or hyperthyroidism. -

Exclusion Criteria:

1. There are communication barriers between researchers and patients.
2. Due to critical condition or unstable vital signs, patients should be transferred to relevant clinical departments for treatment or observation immediately after examination.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received enhanced CT scans via peripheral venous indwelling needle.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
accuracy of prediction model | through study completion, an average of 1 year
  the ratio of correct predictions to the total number of model predictions(%)
the incidence of peripheral venous iodine contrast agent extravasation | One year before and after the prediction model is put into use.
  the number of iodine contrast agent extravasation times divided by the total number of enhanced CT examinations during the same period(%)

CONTACTS AND LOCATIONS:
Overall Officials: Wenyan Zhang, Master, Principal Investigator — Tongji Hospital
Locations (1):
- TongjiHospital, Wuhan, Hubei, China